CLINICAL TRIAL: NCT03992534
Title: Feasibility, Safety, Tolerance and Assessment of LACTIN-V Use in a Cohort of Pregnant Women at Risk of Preterm Birth
Brief Title: The FLIP-1 Study: Vaginal Lactobacillus Supplementation in Women at High Risk of Preterm Birth
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19QC5168
Record Dates: First submitted 2019-05-01; First posted 2019-06-20 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Preterm Labor; Preterm Birth; Preterm Premature Rupture of Membrane; Cervical Incompetence; Miscarriage in Second Trimester; Miscarriage in Third Trimester
Keywords: Pregnancy; Preterm labour; Preterm delivery; Vaginal microbiome; Infection; Next generation sequencing; Lactobacillus
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth; Preterm Premature Rupture of the Membranes; Uterine Cervical Incompetence; Infections | interventions — APF protein, Lactobacillus crispatus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LACTIN-V (Experimental): Name of Product: LACTIN-V (Lactobacillus crispatus CTV-05)
  Dosage: LACTINV is a powder formulation of Lactobacillus crispatus CTV-05 provided in a prefilled vaginal applicator at a dose of 2 x 10^9 CFU of L. crispatus CTV-05. Route of Administration: LACTIN-V powder is administered vaginally using a specially designed applicator.
  Formulation: LACTIN-V is supplied as a pre-filled, single-use applicator. Each applicator contains LACTIN-V powder at a dose of 2 x 10^9 CFU. The LACTIN-V powder formulation contains L. crispatus CTV-05 and a preservation matrix containing inactive excipients of non-animal origin.
  Interventions: Combination Product: LACTIN-V

INTERVENTIONS:
Combination Product: LACTIN-V — Vaginal supplementation with L. crispatus CTV-05.
  Other Names: Lactobacillus crispatus

SUMMARY:
Preterm birth (PTB) is the primary cause of infant death worldwide. It has been shown that a vaginal microbiota deplete in Lactobacillus species is a risk factor for preterm labour. Conversely a vaginal microbiota dominated by Lactobacillus crispatus appears to be protective for these adverse outcomes. A wide range of 'over the counter' Lactobacillus spp. containing products targeted at 'vaginal health' and formulated for vaginal administration are available, but most of them do not contain vaginal species of Lactobacillus. The primary aim of this study is to determine whether vaginal supplementation with L. crispatus CTV-05 is associated with colonisation.

DETAILED DESCRIPTION:
Pregnant women at Queen Charlotte's and Chelsea Hospital and St Mary's Hospital London who are defined as being at a higher than background risk for preterm labour will be recruited into this study. Women at risk of pre-term labour will include those with either previous LLETZ, previous preterm birth, previous second trimester pregnancy loss or a combination of these indications.

As part of this interventional study, subjects will be offered supplementation with L. crispatus CTV-05. The preparation of LACTIN-V is administered vaginally using a specially designed applicator.

The primary aim of this study is to determine whether vaginal supplementation with L. crispatus CTV-05 is associated with colonisation.

ELIGIBILITY:
Inclusion Criteria:

* Women at risk of preterm labour
* Women referred to the prematurity clinic
* Women with previous LLETZ (large loop excision of the transformation zone)
* Women with previous preterm birth
* Women with previous second trimester loss

Exclusion Criteria:

* HIV positive women
* Women who are unable to provide informed consent
* Women aged <18
* Women receiving antibiotic treatment within 1 week of recruitment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants that demonstrate a change in vaginal colonisation during and following LACTIN-V use. | 2-4 years
  Microbiological effects of LACTIN-V by laboratory analysis, next generation sequencing

SECONDARY OUTCOMES:
The number of participants with treatment related adverse events following LACTIN-V supplementation in pregnant women at high risk of preterm birth. | 2-4 years
  Participants will be asked about adverse events during clinical review and the safety profile will be recorded.
The number of patients using LACTIN-V that go on to experience preterm birth, PPROM or cervical shortening. | 2-4 years
  Clinical outcomes of participants will be analysed, in accordance with colonisation results

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Bennett, BSc PhD MD, Principal Investigator — Imperial College London
Locations (1):
- Institute of Reproductive Developmental Biology, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months of study completion
Access Criteria: as study protocol

REFERENCES:
- [Background] MacIntyre DA, Chandiramani M, Lee YS, Kindinger L, Smith A, Angelopoulos N, Lehne B, Arulkumaran S, Brown R, Teoh TG, Holmes E, Nicoholson JK, Marchesi JR, Bennett PR. The vaginal microbiome during pregnancy and the postpartum period in a European population. Sci Rep. 2015 Mar 11;5:8988. doi: 10.1038/srep08988. PMID 25758319
- [Background] Brown RG, Marchesi JR, Lee YS, Smith A, Lehne B, Kindinger LM, Terzidou V, Holmes E, Nicholson JK, Bennett PR, MacIntyre DA. Vaginal dysbiosis increases risk of preterm fetal membrane rupture, neonatal sepsis and is exacerbated by erythromycin. BMC Med. 2018 Jan 24;16(1):9. doi: 10.1186/s12916-017-0999-x. PMID 29361936
- [Background] Kindinger LM, Bennett PR, Lee YS, Marchesi JR, Smith A, Cacciatore S, Holmes E, Nicholson JK, Teoh TG, MacIntyre DA. The interaction between vaginal microbiota, cervical length, and vaginal progesterone treatment for preterm birth risk. Microbiome. 2017 Jan 19;5(1):6. doi: 10.1186/s40168-016-0223-9. PMID 28103952
- [Background] Kindinger LM, MacIntyre DA, Lee YS, Marchesi JR, Smith A, McDonald JA, Terzidou V, Cook JR, Lees C, Israfil-Bayli F, Faiza Y, Toozs-Hobson P, Slack M, Cacciatore S, Holmes E, Nicholson JK, Teoh TG, Bennett PR. Relationship between vaginal microbial dysbiosis, inflammation, and pregnancy outcomes in cervical cerclage. Sci Transl Med. 2016 Aug 3;8(350):350ra102. doi: 10.1126/scitranslmed.aag1026. PMID 27488896
- [Background] Stapleton AE, Au-Yeung M, Hooton TM, Fredricks DN, Roberts PL, Czaja CA, Yarova-Yarovaya Y, Fiedler T, Cox M, Stamm WE. Randomized, placebo-controlled phase 2 trial of a Lactobacillus crispatus probiotic given intravaginally for prevention of recurrent urinary tract infection. Clin Infect Dis. 2011 May;52(10):1212-7. doi: 10.1093/cid/cir183. Epub 2011 Apr 14. PMID 21498386
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435